CLINICAL TRIAL: NCT05182008
Title: A Patient Decision Aid for Method of Early Abortion: a Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other); University of British Columbia (Other); IWK Health Centre (Other)
Responsible Party: Principal Investigator, Melissa Brooks, Obgyn, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NSHA43377
Record Dates: First submitted 2021-12-12; First posted 2022-01-10 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Abortion in First Trimester; Abortion Early; Decision Aid; Clinical Decision-making; Abortion, Therapeutic
Keywords: Abortion; Decision aid
MeSH Terms: interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Decision Aid (Experimental): Patients will be guided to an online interactive decision aid tool.
  Interventions: Other: Decision aid
- Usual Care (Active Comparator): Patients will be guided to visit the clinic website of the Nova Scotia Women's Choice Clinic.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Decision aid — Online interactive decision aid on method of early abortion
  Arms: Decision Aid
Other: Usual care — Patients will be directed to the abortion clinic website
  Arms: Usual Care

SUMMARY:
Introduction: There are two options for women seeking early pregnancy termination in Canada; either surgical or medication abortion. When making a decision about which option is best for them, patient must consider their values as well as social resources and circumstances Patient decision aids (PtDAs) are tools to help patients make health-related decisions, particularly when no 'best' choice exist.

Our research team has developed an online interactive patient decision aid on method of abortion based on international standards for decision aid development. We would like to investigate whether it leads to improved decisional quality in patients seeking early abortion.

Methods: Phase 1 will be development of an abortion knowledge assessment tool. We will start by developing ten multiple choice questions based on information that is classically included in abortion education material. The goal is to ultimately include 5-7 well-performing questions in the trial. The ten questions will be sent to content experts to answer and rate. They will rate the questions on representativeness and importance. The questions will also be administered to community members without specific abortion knowledge. Results will be used to assess content validity and discriminator validity and revise the questionnaire.

Phase 2 will be a randomized trial of people seeking abortion at less than 63 days gestation. Those who wish to participate will be randomized either the decision aid (study group) or the standard abortion clinic website (control). They will then be asked to participate in a survey immediately after they are finished reviewing the decision aid or website to. This survey will include questions about their decision, demographics, medical history, and their level of knowledge about abortion methods (by administering the knowledge assessment tool described above). The evaluation of the decision making will be measured using the Decisional Conflict Score. Four weeks post procedure, participants will be contacted by e-mail again and asked to complete a second survey identifying which type of abortion they underwent along with an inventory of perceived adverse treatment effects, as well as completing a Satisfaction with Decision Scale (SWD)

DETAILED DESCRIPTION:
There are two options for women seeking early pregnancy termination in Canada; either surgical or medication abortion. Each offers unique benefits and drawback. When making a decision about which option is best for them, patient must consider their values as well as social resources and circumstances. These decisions must be made quickly because of the time sensitive nature of abortion. Research has shown that people seeking abortion value making an informed decision on method.

Patient decision aids (PtDAs) are tools to help patients make health-related decisions, particularly when no 'best' choice exist. Research shows that in comparison to usual care, decision aids have been shown to improve patient knowledge and risk perception, reduce decisional conflict, and promote shared decision making and value-congruent decisions (i.e. decisions that are in alignment with the patients stated values and priorities) Our research team has developed an online interactive patient decision aid on method of abortion based on international standards for decision aid development. We would like to investigate whether it leads to improved decisional quality in patients seeking early abortion.

Phase 1 will be development of an abortion knowledge assessment tool. This tool will be used in Phase 2 of the study to evaluate decision quality. We will start by developing ten multiple choice questions based on information that is classically included in abortion education material. The goal is to ultimately include 5-7 well-performing questions in the trial. The ten questions will be sent to content experts to answer and rate. They will rate the questions on representativeness (Overall how well does this question represent key facts that a patient should know before deciding about abortion method?) and importance (How important is this question for patients to understand to be considered informed?). The questions will also be administered to community members without specific abortion knowledge. Based on data from these surveys the questions will be revised. To ensure content validity, only questions the experts rate as sufficiently representative and important will be included. Discriminant validity will be evaluated by comparing the scores of content experts to those of community members. Only questions with adequate discriminant validity will be included. Content experts will be persons known to the primary investigator and will be recruited directly. Community members will be recruited online though social media (eg. Facebook). Both content experts and community members will complete an online consent form and online survey.

Phase 2 of the study will be integrated into the standard workflow of the Nova Scotia Women's Clinic. Patients are able to self refer to the clinic and during the initial intake phone call, they will be asked if they can be contacted by the research coordinator to discuss study participation. Those who agree will be contacted by the research coordinator to review the study and patients will be ask if they would like to participate in the they study. Those who wish to participate will be randomized and e-mailed a weblink to an online consent form and either the decision aid (study group) or the standard NSWCC website (control). Participants will be randomized in a 1:1 ratio within blocks of size 2, 4, and 6 (in random order). To further ensure the randomization is concealed, a statistician who is not on the study team will generate the sequence using the R package, blockrand. They will then be asked to participate in a survey immediately after they are finished reviewing the decision aid or website to. This survey will include questions about their decision, demographic information, medical history,and their level of knowledge about abortion methods (by administering the knowledge assessment tool described above). The evaluation of the decision making will be measured using the Decisional Conflict Score, which measures the quality of the decision making process and consist of question for which patients rate their experiences on a scale of strongly agree or disagree. Four weeks post procedure, participants will be contacted by e-mail again and asked to complete a second survey identifying which type of abortion they underwent along with an inventory of perceived adverse treatment effects, as well as completing a Satisfaction with Decision Scale (SWD)

ELIGIBILITY:
Inclusion Criteria:

* person of reproductive age seeking termination of pregnancy, felt to be within the eligible period for a medication abortion (<9 weeks or 63 days from last menstrual period), can provide consent, has access to internet and a valid email address and be able to read and speak English.

Exclusion Criteria:

* Participants will be excluded from the four week follow up survey if they are subsequently found to be ineligible for medication abortion (pregnancy too advanced or if there are medical contraindications), if they miscarry spontaneously, or choose to continue their pregnancy.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Decisional Conflict Score | Immediately after use of intervention (decision aid) or usual care condition (clinic website)
  The DCS consists of 16 statements that participants rate from "strongly agree" [0] to "strongly disagree" [4]; scores are summed, divided by 16, and multiplied by 25 (for a score out of 100). High scores indicate greater decisional conflict.

SECONDARY OUTCOMES:
Satisfaction with decision score (SWD) | 4 weeks after enrolment (after abortion complete)
  A six-item attitude Likert scale that has been shown to be a reliable and valid measure of patients' satisfaction with their healthcare-related decisions. It is rated on a 1-5 scale (1= strongly disagree; 5 = strongly agree). Higher scores indicate higher satisfaction with decision.
Decision concordance | 4 weeks after enrolment (after abortion complete)
  Decision concordance will be calculated by comparing the stated decision preference at time 0 (for those who express a preference) to the actual method chosen by each patient as measured 4 weeks later. It will be expressed at a percentage.
Knowledge of abortion method score | Immediately after use of intervention (decision aid) or usual care condition (clinic website)
  The knowledge score will be calculated by dividing the number of correct answers by the total number of questions and multiplied by 100 (percentage correct).

OTHER OUTCOMES:
Correlation between SWD scores and patient reported side effects | 4 weeks after enrolment (after abortion complete)
  Patient reported side effect will be measured by a scale created for the study based on the brief pain inventory. This is a Likert scale for patient to rate how side effects interfered with their daily functioning. Higher scores indicate higher levels of interference in activity.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Brooks, Principal Investigator — Dalhousie University
Locations (1):
- QEII Health Sciences Center, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Undecided